CLINICAL TRIAL: NCT06632197
Title: Non-invasive Monitoring of Mixed Venous Oxygen Saturation Using the Capnodynamic Method in Adults
Acronym: CAPNO-SVO2
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Principal Investigator, Isabel Magaña Bru, MD Intesive Care Medicine, Principal Investigator, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Other Study IDs: CAPNO-SVO2
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Ventilatory Failure; Cardiac Failure; Mechanical Ventilation Pressure High
MeSH Terms: conditions — Hypoventilation; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to compare the accuracy and correlation of the capnodynamic method for measuring mixed venous oxygen saturation (SvO2) with the standard reference method (pulmonary artery catheter), with the potential for the capnodynamic method to replace the traditional method in selected cases.

DETAILED DESCRIPTION:
The main objective is to evaluate the accuracy and correlation of mixed venous oxygen saturation (SvO2) measured using the capnodynamic method in comparison with the invasive standard method using co-oximetry with a pulmonary artery catheter (PAC) Swan-Ganz, with the potential to replace it in selected cases, in patients who would benefit from hemodynamic monitoring with PAC for their clinical management and decision-making.

The investigator will also study the following secondary objectives:

* To assess whether the capnodynamic method (Capno-SvO2) detects changes over time in the studied variable (SvO2), showing good concordance and magnitude compared to the reference method.
* To evaluate the progression and trend of the Capno-SvO2 method in different clinical situations, such as in adult respiratory distress syndrome and patients with other respiratory pathologies, as well as patients with cardiac conditions.
* To assess the ability of the Capno-SvO2 method to detect changes in mixed venous oxygen saturation in response to therapeutic interventions (e.g., adjustments in mechanical ventilation, use of inotropes, vasopressors, or fluid therapy) or moderate hemodynamic changes.
* To evaluate the correlation between mixed venous oxygen saturation measured using the Capno-SvO2 method and other hemodynamic parameters, such as cardiac output, central venous pressure, and cardiac index.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Not participating in any other interventional study at the time of the study.
* Patients under controlled mechanical ventilation in passive conditions.
* Situations where the responsible physician deems that, for the benefit of clinical management and therapeutic decision-making, the patient would benefit from the placement of a pulmonary artery catheter (Swan-Ganz) and/or monitoring of central or mixed venous saturation.
* Obtaining informed consent.

Exclusion Criteria:

* Failure to obtain informed consent.
* No need for invasive mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in the ICU of the Hospital Universitario de la Princesa.
  The study population will include all patients with medical conditions (respiratory or cardiac) who could benefit from the placement of a PAC and/or the monitoring of mixed venous saturation for clinical management and decision-making, or monitoring of central venous saturation if a pulmonary artery catheter is not required.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Mixed venous oxygen saturation (SvO2) | 24 hours
  measured using the capnodynamic method in comparison with the invasive standard method using co-oximetry with a pulmonary artery catheter (PAC).

SECONDARY OUTCOMES:
Cardiac output | 24 hours
  measured using the capnodynamic method in comparison with the invasive standard method using co-oximetry with a pulmonary artery catheter (PAC).